CLINICAL TRIAL: NCT03788980
Title: Risk Factors for Complications After Carotid Endarterectomy: A Multicenter International Observational Study
Brief Title: Risk Factors for Complications After Carotid Endarterectomy
Status: Terminated | Type: Observational
Why Stopped: Lack of funding and resources
Sponsor: Ohio State University (Other)
Collaborators: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Sponsor
Other Study IDs: 2018H0044
Record Dates: First submitted 2018-12-26; First posted 2018-12-28 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Complications; Postoperative Cognitive Dysfunction
Keywords: Endarterectomy
MeSH Terms: conditions — Postoperative Complications; Postoperative Cognitive Complications | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- carotid endarterectomy group: patients undergoing carotid endarterectomy
  Interventions: Procedure: Carotid endarterectomy; Diagnostic Test: Mini Mental Status Examination

INTERVENTIONS:
Procedure: Carotid endarterectomy — Patients will undergo a surgery called carotid endarterectomy where a surgeon will remove material that causes carotid stenosis (i.e. plaque)
  Other Names: CAE
Diagnostic Test: Mini Mental Status Examination — Short questionnaire used to diagnose cognitive dysfunction
  Other Names: MMSE

SUMMARY:
This study may determine the incidence of complications that occur after patients undergo a surgery called Carotid Endarterectomy (CEA), which is a surgery that aims to decrease the risk of strokes in patients with a condition called carotid stenosis. Medical records will be accessed to find any information pertaining to postoperative complications. Additionally, it may determine the cognitive dysfunction of patients undergoing CEA, assessed by Mini Mental Status Examination (MMSE).

DETAILED DESCRIPTION:
This is a multicenter prospective observational study; data will be collected from two sites: the lead site in Columbus, Ohio, USA and an international site in Girona, Spain for a total of 354 patients. The objective of this study is to determine the incidence of complications that occur after patients undergo a surgery called Carotid Endarterectomy (CEA), which is a surgery that aims to decrease the risk of strokes in patients with a condition called carotid stenosis. Patients who undergo CEA are at increased risk of cardiovascular complications because of the high incidence of coexisting heart disease, high blood pressure, and diabetes. Common complications that occur after CEA are wound hematoma (collection of blood at the wound) and intracerebral hemorrhage (bleeding in the brain). Medical records will be accessed to find any information pertaining to postoperative complications. Another objective of this study is to determine the cognitive dysfunction of patients undergoing CEA. This will be measured by a Mini Mental Status Examination (MMSE) which will occur in person before the surgery and 30 days after the surgery over the phone. This study may provide data that will help identify how to optimize recovery for future CEA patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients males or females, 18 years of age and older
* Scheduled to undergo Carotid Endarterectomy

Exclusion Criteria:

1. Pregnant women
2. Incarcerated individuals
3. Patients not able to consent for themselves
4. Any disease or condition deemed by the investigator to disqualify the patient
5. Participating in any interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older scheduled to undergo carotid endarterectomy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Complication rate | 30 days
  Incidence of postoperative complications and identify the associated risk factors.

SECONDARY OUTCOMES:
Cognitive Dysfunction | 30 days
  the incidence of cognitive dysfunction based on Mini Mental Status Examination

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Bergese, MD, Principal Investigator — The Ohio State University Wexner Medical Center Department of Anesthesiology
Locations (2):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States
- Hospital Universitari de Girona Dr. Josep Trueta, Girona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
The de-identified date from the international site and the data collected at the main site will be analyzed at The Ohio State University Wexner Medical Center.

REFERENCES:
- [Background] Endarterectomy for asymptomatic carotid artery stenosis. Executive Committee for the Asymptomatic Carotid Atherosclerosis Study. JAMA. 1995 May 10;273(18):1421-8. PMID 7723155
- [Background] Stoneham MD, Thompson JP. Arterial pressure management and carotid endarterectomy. Br J Anaesth. 2009 Apr;102(4):442-52. doi: 10.1093/bja/aep012. Epub 2009 Feb 20. PMID 19233880
- [Background] McCollum PT, da Silva A, Ridler BD, de Cossart L. Carotid endarterectomy in the U.K. and Ireland: audit of 30-day outcome. The Audit Committee for the Vascular Surgical Society. Eur J Vasc Endovasc Surg. 1997 Nov;14(5):386-91. doi: 10.1016/s1078-5884(97)80289-4. PMID 9413380
- [Background] Ferguson GG, Eliasziw M, Barr HW, Clagett GP, Barnes RW, Wallace MC, Taylor DW, Haynes RB, Finan JW, Hachinski VC, Barnett HJ. The North American Symptomatic Carotid Endarterectomy Trial : surgical results in 1415 patients. Stroke. 1999 Sep;30(9):1751-8. doi: 10.1161/01.str.30.9.1751. PMID 10471419
- [Background] Robinson TG, James M, Youde J, Panerai R, Potter J. Cardiac baroreceptor sensitivity is impaired after acute stroke. Stroke. 1997 Sep;28(9):1671-6. doi: 10.1161/01.str.28.9.1671. PMID 9303008
- [Background] Rothwell PM, Giles MF, Chandratheva A, Marquardt L, Geraghty O, Redgrave JN, Lovelock CE, Binney LE, Bull LM, Cuthbertson FC, Welch SJ, Bosch S, Alexander FC, Silver LE, Gutnikov SA, Mehta Z; Early use of Existing Preventive Strategies for Stroke (EXPRESS) study. Effect of urgent treatment of transient ischaemic attack and minor stroke on early recurrent stroke (EXPRESS study): a prospective population-based sequential comparison. Lancet. 2007 Oct 20;370(9596):1432-42. doi: 10.1016/S0140-6736(07)61448-2. PMID 17928046
- [Background] Asiddao CB, Donegan JH, Whitesell RC, Kalbfleisch JH. Factors associated with perioperative complications during carotid endarterectomy. Anesth Analg. 1982 Aug;61(8):631-7. PMID 7201265
- [Background] Kunkel JM, Gomez ER, Spebar MJ, Delgado RJ, Jarstfer BS, Collins GJ. Wound hematomas after carotid endarterectomy. Am J Surg. 1984 Dec;148(6):844-7. doi: 10.1016/0002-9610(84)90451-3. PMID 6507761
- [Background] Karapanayiotides T, Meuli R, Devuyst G, Piechowski-Jozwiak B, Dewarrat A, Ruchat P, Von Segesser L, Bogousslavsky J. Postcarotid endarterectomy hyperperfusion or reperfusion syndrome. Stroke. 2005 Jan;36(1):21-6. doi: 10.1161/01.STR.0000149946.86087.e5. Epub 2004 Dec 2. PMID 15576656
- [Background] Naylor AR, Evans J, Thompson MM, London NJ, Abbott RJ, Cherryman G, Bell PR. Seizures after carotid endarterectomy: hyperperfusion, dysautoregulation or hypertensive encephalopathy? Eur J Vasc Endovasc Surg. 2003 Jul;26(1):39-44. doi: 10.1053/ejvs.2002.1925. PMID 12819646
- [Background] Russell DA, Gough MJ. Intracerebral haemorrhage following carotid endarterectomy. Eur J Vasc Endovasc Surg. 2004 Aug;28(2):115-23. doi: 10.1016/j.ejvs.2004.03.020. PMID 15234690
- [Background] Nordlander M, Sjoquist PO, Ericsson H, Ryden L. Pharmacodynamic, pharmacokinetic and clinical effects of clevidipine, an ultrashort-acting calcium antagonist for rapid blood pressure control. Cardiovasc Drug Rev. 2004 Fall;22(3):227-50. doi: 10.1111/j.1527-3466.2004.tb00143.x. PMID 15492770
- [Background] Aronson S, Dyke CM, Stierer KA, Levy JH, Cheung AT, Lumb PD, Kereiakes DJ, Newman MF. The ECLIPSE trials: comparative studies of clevidipine to nitroglycerin, sodium nitroprusside, and nicardipine for acute hypertension treatment in cardiac surgery patients. Anesth Analg. 2008 Oct;107(4):1110-21. doi: 10.1213/ane.0b013e31818240db. PMID 18806012
- [Background] Singla N, Warltier DC, Gandhi SD, Lumb PD, Sladen RN, Aronson S, Newman MF, Corwin HL; ESCAPE-2 Study Group. Treatment of acute postoperative hypertension in cardiac surgery patients: an efficacy study of clevidipine assessing its postoperative antihypertensive effect in cardiac surgery-2 (ESCAPE-2), a randomized, double-blind, placebo-controlled trial. Anesth Analg. 2008 Jul;107(1):59-67. doi: 10.1213/ane.0b013e3181732e53. PMID 18635468
- [Background] Ericsson H, Bredberg U, Eriksson U, Jolin-Mellgard A, Nordlander M, Regardh CG. Pharmacokinetics and arteriovenous differences in clevidipine concentration following a short- and a long-term intravenous infusion in healthy volunteers. Anesthesiology. 2000 Apr;92(4):993-1001. doi: 10.1097/00000542-200004000-00016. PMID 10754618
- [Background] Muller L, Bobbia X, Toumi M, Louart G, Molinari N, Ragonnet B, Quintard H, Leone M, Zoric L, Lefrant JY; AzuRea group. Respiratory variations of inferior vena cava diameter to predict fluid responsiveness in spontaneously breathing patients with acute circulatory failure: need for a cautious use. Crit Care. 2012 Oct 8;16(5):R188. doi: 10.1186/cc11672. PMID 23043910